CLINICAL TRIAL: NCT00680849
Title: Enhancing Support for Women With Type 2 Diabetes: Follow-Up
Status: Completed | Type: Observational
Sponsor: Oregon Research Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HL077120
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Coronary Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Treatment condition from first study. This is a follow-up study.
- 2: Control condition from first study.

SUMMARY:
This study is a 5-year continuation of "The Mediterranean Lifestyle Program." The purpose of this follow-up study is to determine the long-term effects from prior participation in an intervention promoting healthful eating, exercise, quitting smoking, stress management, and social support. Participants are post-menopausal women with type 2 diabetes.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is the leading cause of death and functional limitations among women in the U.S. Postmenopausal women with diabetes are at especially high risk of CHD, but CHD research with this population is very limited. This project addresses the poorly understood "natural history" of long-term maintenance of change in multiple behaviors (i.e., dietary, physical activity, social support, smoking cessation, and stress management) related to CHD risk, as well as the effects of theoretically important mediating variables on relapse and maintenance. The study is a continuation of a research project that has already demonstrated significant and consistent positive effects of a lifestyle change intervention on reduction of behavioral CHD risk factors. This research relies on a framework that synthesizes social-cognitive, social-ecologic, and goal-systems theories.

ELIGIBILITY:
Inclusion Criteria: All participants in the original study are eligible. The inclusion criteria for the original study were:

* diagnosis of type 2 diabetes for at least 6 months
* being post-menopausal
* living independently (e.g., not in an institution or nursing home)
* having a telephone
* ability to read English
* not being developmentally disabled, and
* living within 30 miles of the Eugene-Springfield metropolitan area.

Exclusion Criteria: Exclusion criteria for the original study included:

* being older than 75 years of age
* having life-threatening illnesses, or
* planning to move from the local area within the time span of the study.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in prior study: Enhancing Support for Women With Type 2 Diabetes, "The Mediterranean Lifestyle Program."
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2003-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Food Frequency Questionnaire for Fruits, Vegetables and percent calories from fat (FFQ) by Kristal and colleagues | annually, 36 months - 84 months

SECONDARY OUTCOMES:
Lipids, weight loss | annually, 36 months - 84 months

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J. Toobert, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Background] Barrera M Jr, Toobert DJ, Angell KL, Glasgow RE, Mackinnon DP. Social support and social-ecological resources as mediators of lifestyle intervention effects for type 2 diabetes. J Health Psychol. 2006 May;11(3):483-95. doi: 10.1177/1359105306063321. PMID 16774900
- [Background] Barrera M, Strycker LA, Mackinnon DP, Toobert DJ. Social-ecological resources as mediators of two-year diet and physical activity outcomes in type 2 diabetes patients. Health Psychol. 2008 Mar;27(2S):S118-25. doi: 10.1037/0278-6133.27.2(Suppl.).S118. PMID 18377153
- [Background] Greene GW, Nebeling LC, Greaney ML, Lindsay AC, Hardwick CK, Toobert DJ, Resnicow K, Williams GC, Elliot DL, Goldman Sher T, McGregor HA, Domas A, DeFrancesco CA, Peterson KE. A qualitative study of a nutrition working group. Health Promot Pract. 2007 Jul;8(3):299-306. doi: 10.1177/1524839906292587. Epub 2007 May 23. PMID 17522413
- [Background] Hellsten LA, Nigg C, Norman G, Burbank P, Braun L, Breger R, Coday M, Elliot D, Garber C, Greaney M, Lees F, Matthews C, Moe E, Resnick B, Riebe D, Rossi J, Toobert D, Wang T. Accumulation of behavioral validation evidence for physical activity stage of change. Health Psychol. 2008 Jan;27(1S):S43-53. doi: 10.1037/0278-6133.27.1(Suppl.).S43. PMID 18248105
- [Background] King AC, Toobert D, Ahn D, Resnicow K, Coday M, Riebe D, Garber CE, Hurtz S, Morton J, Sallis JF. Perceived environments as physical activity correlates and moderators of intervention in five studies. Am J Health Promot. 2006 Sep-Oct;21(1):24-35. doi: 10.1177/089011710602100106. PMID 16977910
- [Background] Ritzwoller DP, Toobert D, Sukhanova A, Glasgow RE. Economic analysis of the Mediterranean Lifestyle Program for postmenopausal women with diabetes. Diabetes Educ. 2006 Sep-Oct;32(5):761-9. doi: 10.1177/0145721706291757. PMID 16971709
- [Background] Strycker LA, Duncan SC, Chaumeton NR, Duncan TE, Toobert DJ. Reliability of pedometer data in samples of youth and older women. Int J Behav Nutr Phys Act. 2007 Feb 17;4:4. doi: 10.1186/1479-5868-4-4. PMID 17306031
- [Background] Toobert DJ, Glasgow RE, Strycker LA, Barrera M Jr, Ritzwoller DP, Weidner G. Long-term effects of the Mediterranean lifestyle program: a randomized clinical trial for postmenopausal women with type 2 diabetes. Int J Behav Nutr Phys Act. 2007 Jan 17;4:1. doi: 10.1186/1479-5868-4-1. PMID 17229325